CLINICAL TRIAL: NCT00788814
Title: Women Physical Disability and Depression: Communities Responding Now!
Brief Title: Study of Pathways Curriculum for Use With WPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland State University (Other)
Responsible Party: Principal Investigator, Dena Hassouneh, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH079818-01A1 (NIH); 1R01MH079818-01A1 (NIH)
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control (Other): Control group
  Interventions: Behavioral: Pathways

INTERVENTIONS:
Behavioral: Pathways — Strength-based curriculum addressing depression in women with with physical disabilities

SUMMARY:
Study to assess the efficacy of a modified Pathways curriculum in treating depressive symptoms in women with physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Women with physical disability requiring accommodation for major mobility limitations
* CES-D score of 16 or higher -

Exclusion Criteria:

* Active suicidality
* Diagnosis of Schizophrenia, Schizoaffective D/O, Psychosis NOS
* Currently receiving other psychotherapy -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | pre-test, post-test weeks, 12, 18, 24

CONTACTS AND LOCATIONS:
Overall Officials: Dena M Hassouneh, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States